CLINICAL TRIAL: NCT00630864
Title: The Effects of Fx-1006A on Transthyretin Stabilization and Clinical Outcome Measures in Patients With Non-V30M Transthyretin Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX1A-201; B3461022
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Transthyretin-associated Amyloidosis With Polyneuropathy
Keywords: Transthyretin, TTR, amyloidosis, TTR amyloidosis, polyneuropathy
MeSH Terms: conditions — Amyloidosis; Polyneuropathies | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Fx-1006A 20mg soft gelatin capsules once daily for 12 months
  Interventions: Drug: Fx-1006A

INTERVENTIONS:
Drug: Fx-1006A — During Part 1, patients will receive Fx-1006A 20mg soft gelatin capsules once daily (at the same time each day) for two weeks. During Part 2, patients will receive Fx-1006A 20mg soft gelatin capsules once daily to complete a total of 12 months of dosing

SUMMARY:
This is an open-label, multicenter, international study designed to determine TTR stabilization as well as Fx-1006A safety and tolerability, and its effects on clinical outcomes in patients with non-V30M TTR amyloidosis.

Strong pre-clinical and clinical evidence support a daily dose of 20 mg of Fx-1006A to be the optimum dose to achieve stabilization of tetrameric TTR in ATTR-PN patients. Since disease presentation is similar between V30M and non-V30M TTR mutations associated with ATTR-PN and Fx-1006A has been shown to stabilize wild-type and V30M TTR in vitro and ex vivo, the present study is being conducted to determine the effects of Fx-1006A on TTR stabilization in ATTR-PN patients with TTR mutations other than V30M. Safety and exploratory efficacy of Fx-1006A administered once daily for 12 months will also be evaluated in this patient population.

This is an open-label, multicenter, international study designed to determine TTR stabilization as well as Fx-1006A safety and tolerability, and its effects on clinical outcomes in patients with non-V30M TTR amyloidosis. The study will be conducted in two parts. Part 1 will include a six-week dosing period during which all enrolled patients will receive oral Fx-1006A 20 mg soft gelatin capsules once daily for six weeks. At Week 6, blood samples will be collected from each patient to determine TTR stabilization. Patients who complete the Week 6 visit will continue receiving daily oral Fx-1006A 20 mg for up to a total of 12 months during Part 2 of this study. If it is determined that a patient is not stabilized at Week 6, the patient will be discontinued from the study.

During Part 2, clinical outcomes will be measured at Months 6 and 12, based on NIS, Norfolk QOL-DN, mBMI, NCS, HRDB, SF-36, Karnofsky score, and echocardiography; NT-pro-BNP and troponin I levels will be measured at Baseline, Weeks 2 and 6, and Months 3, 6, and 12.

Pharmacokinetic measurements will be made using samples collected at Baseline, Week 6, and Months 6 and 12.

Safety and tolerability will be assessed throughout the study based on vital signs, physical examinations, ECG, echocardiography, 24-hour Holter monitoring, clinical laboratory tests (hematology, serum chemistry, and urinalysis), and monitoring adverse events and concomitant medication use.

Day 1 will be defined as administration of the first dose of study drug. Clinic Visits will be conducted during Screening (Days -30 to -1) and at Baseline (Day 0), and Week 2, and Week 6, and Months 3, 6, and 12 (± 2 weeks of the scheduled date for post-Baseline visits). Monthly telephone contacts (+ 1 week of the scheduled date) will be made during months in which no investigative site visits are scheduled (Months 4, 5, 7, 8, 9, 10, and 11) for assessment of adverse events and concomitant medications. A final telephone contact to assess adverse events and concomitant medication usage will be made 30 days after the last dose of study drug.

Patients who discontinue from the study at any time following enrollment will have a final visit performed, including all safety assessments, at the time of discontinuation. Any patient discontinuing after the Month 6 visit will also have all exploratory assessments performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient has amyloid documented by biopsy (in accordance with institutional site standard of care).
* Patient has documentation of one of the following targeted TTR mutations: Ser77Tyr, Thr60Ala, Tyr114Cys, Leu58His, Glu89Gln, Ser77Phe, Thr49Ala, Ile107Val, Val30Ala, Gly47Ala, Gly47Glu, Leu55Arg, Lys70Asn, Ile84Thr, Ile107Met. Patients with mutations other than those listed may be enrolled only after approval by the Sponsor.
* Patient has peripheral and/or autonomic neuropathy and/or cardiomyopathy with a Karnofsky Performance Status ≥ 50.
* Patient is aged ≥18 to 75 years, inclusive.
* If female, patient is post-menopausal, surgically sterilized, or willing to use two acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide) throughout the study and for 3 months from the end of the study. (A condom alone is not considered an acceptable method of birth control.) If male with a female partner of childbearing potential, willing to use two acceptable methods of birth control for the duration of the study. For both females and males, acceptable birth control must be used for at least 3 months after the last dose of study medication.
* Patient is, in the opinion of the investigator, willing and able to comply with the study medication regimen and all other study requirements.

Exclusion Criteria:

* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs), defined as greater than 3-4 times/month (ibuprofen and nimesulide will be permitted).
* Patient has primary or secondary amyloidosis.
* Patient has TTR-associated amyloidosis with V30M mutation.
* If female, patient is pregnant or breast feeding.
* Patient has received prior liver transplantation.
* Patient is expected to undergo liver transplantation within 12 months after enrollment.
* Patient with positive results for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), and/or human immunodeficiency virus (HIV).
* Patient has renal insufficiency (creatinine clearance < 30 ml/min).
* Patient has liver function test abnormalities: alanine transaminases (ALT) and/or aspartate transaminases (AST) > 2 times upper limit of normal (ULN) that in the medical judgment of the investigator are due to reduced liver function or active liver disease.
* Patient has a New York Heart Association (NYHA) Functional Classification ≥ III.
* Patient has other causes of sensorimotor neuropathy (B12 deficiency, Diabetes Mellitus, HIV treated with retroviral medications, thyroid disorders, alcohol abuse, and chronic inflammatory diseases).
* Patient has prior non-amyloid cardiac disease such as: myocardial infarction due to obstructive coronary artery disease, active non-amyloid cardiomyopathy (e.g., symptomatic left ventricular dysfunction from any cause other than amyloid, patients with a primary diagnosis of symptomatic valvular heart disease)
* Patient has a co-morbidity anticipated to limit survival to less than 12 months.
* Patient has received an investigational drug/device and/or participated in another clinical investigational study within 60 days before Baseline (Day 0).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Johns Hopkins Hospital, Baltimore, Maryland, United States
- CHU de Bicetre, Paris, France
- Universitatsklinikum Munster, Transplant Hepatology, Münster, Germany
- Centro per lo Studio e la Cura delle Amiloidosi Sistemiche, Irccs - Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Derived] Merlini G, Coelho T, Waddington Cruz M, Li H, Stewart M, Ebede B. Evaluation of Mortality During Long-Term Treatment with Tafamidis for Transthyretin Amyloidosis with Polyneuropathy: Clinical Trial Results up to 8.5 Years. Neurol Ther. 2020 Jun;9(1):105-115. doi: 10.1007/s40120-020-00180-w. Epub 2020 Feb 27. PMID 32107748
- [Derived] Huber P, Flynn A, Sultan MB, Li H, Rill D, Ebede B, Gundapaneni B, Schwartz JH. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. Amyloid. 2019 Dec;26(4):203-209. doi: 10.1080/13506129.2019.1643714. Epub 2019 Jul 27. PMID 31353964
- [Derived] Gundapaneni BK, Sultan MB, Keohane DJ, Schwartz JH. Tafamidis delays neurological progression comparably across Val30Met and non-Val30Met genotypes in transthyretin familial amyloid polyneuropathy. Eur J Neurol. 2018 Mar;25(3):464-468. doi: 10.1111/ene.13510. Epub 2017 Dec 26. PMID 29115008
- [Derived] Merlini G, Plante-Bordeneuve V, Judge DP, Schmidt H, Obici L, Perlini S, Packman J, Tripp T, Grogan DR. Effects of tafamidis on transthyretin stabilization and clinical outcomes in patients with non-Val30Met transthyretin amyloidosis. J Cardiovasc Transl Res. 2013 Dec;6(6):1011-20. doi: 10.1007/s12265-013-9512-x. Epub 2013 Oct 8. PMID 24101373

RESULTS

PARTICIPANT FLOW:
Groups:
- Tafamidis: Participants with transthyretin (TTR) variants other than valine replaced by methionine at position 30 (V30M) received tafamidis (Fx-1006A) 20 milligram (mg) capsule orally once daily up to Week 6 in Part 1, participants who achieved TTR stabilization at Week 6 or as per investigator's discretion continued to receive tafamidis (Fx-1006A) 20 mg capsule orally once daily up to Month 12 in Part 2.
Period: Part 1 (up to Week 6)
Arm/Group | Tafamidis
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1
Period: Part 2 (After Week 6 up to Month 12)
Arm/Group | Tafamidis
Started | 20
Completed | 18
Not Completed | 2
Not completed — Liver transplant | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 63.10 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR) Tetramer at Week 6
Description: TTR tetramer was assessed using a validated immunoturbidimetric assay. The Fraction of Initial (FOI) is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI.
Time Frame: Week 6
Population: Intent-to-Treat (ITT) population included all participants who received at least 1 dose of study medication. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 19
percentage of participants | 94.7 [74.0 to 99.9]

2. Secondary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR) Tetramer at Month 6 and 12
Description: TTR tetramer was assessed using a validated immunoturbidimetric assay. The FOI is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI.
Time Frame: Month 6, Month 12
Population: ITT population included all participants who received at least 1 dose of study medication. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
percentage of participants
  Month 6 (n= 18) | 100.0 [81.5 to 100.0]
  Month 12 (n= 17) | 100.0 [80.5 to 100.0]

3. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after the last dose
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
participants | 17

4. Other Pre Specified Outcome: Number of Participants With Greater Than or Equal to Grade 3 Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. On the basis of intensity, grade 3 was referred as severe, grade 4 as life-threatening and grade 5 as death.
Time Frame: Baseline up to 30 days after the last dose
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
participants | 3

5. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-Emergent Echocardiography (ECHO) Findings
Description: ECHO: investigator assessed test to assess cardiac function. ECHO abnormality criteria: any abnormality, valvular abnormality, pericardial effusion, abnormal regional wall motion, inferior vena cava respiratory variation, posterior (P) left ventricular (LV) wall/septal (S) thickness, right ventricular thickness, ejection fraction, ratio of early (E) diastolic transmitral flow and atrial(A) contraction velocity (E/A), ratio of 'E'to lateral/septal mitral annular velocity (e') (E/e'prime lateral, E/e'prime septal), E deceleration time (DT), isovolumic relaxation time (IVRT).
Time Frame: Day 1 up to Month 12
Population: ITT population. The 'n' for any post-dose incidence included participants with baseline values that were not abnormal (that is treatment-emergent abnormalities). Abnormalities at early termination were excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
participants
  Any ECHO abnormalities (n= 19) | 12
  Pericardial effusion (n= 19) | 2
  Valvular abnormalities- thickening (n= 5) | 3
  Valvular abnormalities - regurgitation (n= 9) | 2
  Abnormal regional wall motion (n= 11) | 2
  Inferior vena cava respiratory variation (n= 13) | 0
  LV P wall thickness >=13 millimeter (mm) (n= 3) | 2
  LV S thickness >=13 mm (n= 3) | 1
  Right ventricular thickness >=7 mm (n= 13) | 6
  E/A ratio >=2 (n= 16) | 3
  E/e'prime Lateral >15 (n= 15) | 3
  E/e'prime Septal >15 (n= 10) | 2
  Ejection fraction < 50 percent (%) (n= 17) | 2
  EDT <= 150 milliseconds (msec) (n= 14) | 1
  IVRT <=70 msec (n= 13) | 2

6. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-Emergent Electrocardiogram (ECG) Findings
Description: ECG: investigator assessed test to assess cardiac function. ECG abnormality criteria: any abnormality, arrhythmia, rhythm, conduction, morphology, myocardial infarction, ST segment, T waves and abnormal U waves.
Time Frame: Day 1 up to Month 12
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
participants
  Any ECG abnormalities (n= 21) | 9
  Arrhythmia (n= 18) | 8
  Rhythm (n= 18) | 1
  Conduction (n= 8) | 2
  Morphology (n= 20) | 0
  Myocardial infarction (n= 18) | 0
  ST segment (n= 20) | 1
  T waves (n=18) | 1
  Abnormal U waves (n= 21) | 0

7. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-Emergent Holter Monitoring Findings
Description: Holter monitoring recorded heart rhythm. Holter monitoring abnormality criteria: any abnormality, atrial fibrillation/flutter, atrial tachycardia, non-sustained ventricular tachycardia (VT), sustained VT and sinus pause.
Time Frame: Day 1 up to Month 12
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
participants
  Any Holter monitoring abnormalities (n= 19) | 9
  Atrial fibrillation/flutter (n= 18) | 1
  Atrial tachycardia (n= 9) | 4
  Non-sustained VT <30 beats (n= 11) | 4
  Sustained VT >=30 beats (n= 19) | 0
  Sinus pause (n= 18) | 1

8. Other Pre Specified Outcome: Number of Participants Who Discontinued Due to Clinical or Laboratory Adverse Events
Time Frame: Baseline up to Month 12
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
participants | 1

9. Other Pre Specified Outcome: Change From Baseline in the Neuropathy Impairment Score (NIS) at Month 6, Month 12
Description: NIS assessed cranial nerves(nerve 3,6; facial, palate and tongue weakness),muscle weakness (respiratory; neck, elbow(E), wrist(W), finger(F), hip, knee(K) flexion; shoulder, thumb abduction; brachioradialis; E, W, hip, K extension; F spread; toe, dorsal and plantar ankle flexors; toe extensors); score: 0-4, higher score=more weakness, reflexes(biceps and triceps brachii; brachioradialis; quadriceps femoris; triceps surae), index F and great toe sensation(touch pressure, pin-prick, vibration, joint position)score:0=normal,1=decreased or 2=absent. Total score=0-244, higher score=more impairment.
Time Frame: Baseline, Month 6, Month 12
Population: ITT population included all participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were analyzed for the specific category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
units on a scale
  Baseline (n= 21) | 48.70 (44.31)
  Change at Month 6 (n= 17) | 2.00 (9.52)
  Change at Month 12 (n= 18) | 5.30 (12.62)

10. Other Pre Specified Outcome: Change From Baseline in the Neuropathy Impairment Score-Lower Limb (NIS-LL) at Month 6, Month 12
Description: NIS-LL: assessed muscle weakness, reflexes and sensation; scored separately for left and right limbs. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) are scored on 0 to 4 scale, higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) were scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS-LL score range 0-88, higher score=greater impairment.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
units on a scale
  Baseline (n= 21) | 27.60 (24.67)
  Change at Month 6 (n= 19) | -0.50 (5.73)
  Change at Month 12 (n= 18) | 2.70 (6.21)

11. Other Pre Specified Outcome: Percentage of Participants With Response to Treatment as Measured by Neuropathy Impairment Score - Lower Limb (NIS-LL) at Month 6, Month 12
Description: Response to treatment was indicated by either improvement (decrease from baseline) or stabilization (change from baseline of 0 to less than [<] 2) in Neuropathy Impairment Score- Lower Limb (NIS-LL) score, based on mean of 2 scores in 1 week period. NIS-LL: assessed muscle weakness, reflexes, sensation. Each item scored separately for left, right limbs. Components of muscle weakness scored on 0(normal) to 4(paralysis) scale, higher score=greater weakness. Components of reflexes, sensation scored 0=normal, 1=decreased, or 2=absent. Total NIS-LL score range 0-88, higher score=greater impairment.
Time Frame: Month 6, Month 12
Population: Data on NIS-LL was reported in individual participant listings but responder status was not statistically summarized.
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Change From Baseline in Total Quality of Life (TQOL) Score at Month 6, Month 12
Description: TQOL= sum of all Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QOL-DN) items,a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on QOL of participants with DN; Item 1 to 7: related to symptoms and presence of symptom was assessed as 1 and absence was assessed as 0. Item 8-35: related to activities of daily living and scored on a 5-point Likert scale, where 0= no problem and 4= severe problem (except item 32, where -2= much better, 0=about the same, 2=much worse). Total TQOL score=-2 to 138;higher score=worse quality of life.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
units on a scale
  Baseline (n= 21) | 47.80 (35.14)
  Change at Month 6 (n= 19) | -4.30 (13.25)
  Change at Month 12 (n= 18) | 0.10 (18.01)

13. Other Pre Specified Outcome: Change From Baseline in Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) Domain Scores at Month 6, Month 12
Description: Norfolk QOL-DN:35-item participant-rated questionnaire to assess impact of DN on QOL; Item 1-7: scored as 1=symptom present, 0=symptom absent. Item 8-35: scored on 5-point Likert scale:0=no problem, 4=severe problem(except item 32: -2=much better, 0=about same, 2=much worse).Norfolk QOL-DN summarized in 5 domains (score range): physical functioning/large fiber neuropathy(-2 to 58), activities of daily living(ADLs) (0 to 20), symptom(0 to 32), small fiber neuropathy(0 to 16), autonomic neuropathy(0 to 12);higher score=greater impairment, for each. Total score=-2 to 138 (higher score=worse QOL).
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
units on a scale
  Physical (P)functioning/large fiber:Baseline(n=21) | 25.60 (18.50)
  P functioning/large fiber: Change at Month 6(n=19) | -2.60 (8.66)
  P functioning/large fiber:Change at Month 12(n=18) | -1.40 (11.71)
  ADLs: Baseline (n=21) | 7.30 (7.01)
  ADLs: Change at Month 6 (n=19) | 0.10 (3.07)
  ADLs: Change at Month 12 (n=18) | 0.90 (2.58)
  Symptoms: Baseline (n=21) | 9.00 (7.50)
  Symptoms: Change at Month 6 (n=19) | -0.90 (3.05)
  Symptoms: Change at Month 12 (n=18) | -0.10 (4.28)
  Small fiber neuropathy (SFN): Baseline (n=21) | 3.90 (4.92)
  SFN: Change at Month 6 (n=19) | -0.30 (2.54)
  SFN: Change at Month 12 (n=18) | 0.70 (3.22)
  Autonomic neuropathy (AN): Baseline (n=21)) | 2.00 (1.96)
  AN: Change at Month 6 (n=19) | -0.50 (1.61)
  AN: Change at Month 12 (n=18) | -0.10 (1.13)

14. Other Pre Specified Outcome: Change From Baseline in Nerve Conduction Studies (NCS) at Month 6, Month 12
Description: NCS: quantitative measures of peripheral nerve dysfunction consists of 5 attributes: peroneal nerve (PN) motor distal latency, PN compound muscle action potential, PN motor conduction velocity, tibial nerve distal motor latency, sural nerve sensory nerve action potential. Normal deviates (Z-score) summated into composite score (higher score=worsened nerve fiber function). Z-score is the defined position of the result in normal probability distribution with a mean of 0 and standard deviation (std) of 1 and describes how far a score is (in std) from the mean.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
Z-score
  Baseline (n= 21) | 6.10 (5.90)
  Change at Month 6 (n= 19) | 0.60 (2.69)
  Change at Month 12 (n= 18) | 0.20 (3.30)

15. Other Pre Specified Outcome: Change From Baseline in Heart Rate Response to Deep Breathing (HRDB) at Month 6 and Month 12
Description: HRDB test was used to evaluate the cardio-vagal response. Participant took a series of 8 deep breaths and average heart rate difference was measured and compared to normative data. The main factor affecting HRDB is age, with older patients showing less heart rate variability. R-R (time between two consecutive R waves in the electrocardiogram) response to deep breathing was reported as the normal deviates (Z-score), the defined position of the result in normal probability distribution with a mean of 0 and standard deviation (std) of 1 and describes how far a score is (in std) from the mean.
Time Frame: Baseline, Month 6, Month 12
Population: ITT population included all participants who received at least 1 dose of study medication. Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were analyzed for the specific category.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Tafamidis
Number analyzed (Participants) | 12
Z-score
  Baseline (n= 12) | -0.70 (2.17)
  Change at Month 6 (n= 6) | 0.00 (2.26)
  Change at Month 12 (n= 7) | -0.1 (1.36)

16. Other Pre Specified Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Month 6, Month 12
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2). mBMI was calculated by multiplying BMI by serum albumin levels [gram/liter (g/L)]. mBMI was measured as kg/m^2*g/L. A progressive decline in mBMI indicated worsening of disease severity.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: kg/m^2*g/L
Arm/Group | Tafamidis
Number analyzed (Participants) | 20
kg/m^2*g/L
  Baseline (n= 20) | 1052.50 (206.66)
  Change at Month 6 (n= 17) | -22.40 (77.01)
  Change at Month 12 (n= 16) | 16.60 (89.33)

17. Other Pre Specified Outcome: Change From Baseline in Overall Quality of Life and Individual Domains of the Short-form-36 (SF-36) at Month 6, Month 12
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health and two total scores (physical component summary [PCS] and mental component summary [MCS]. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
units on a scale
  PCS: Baseline (n= 21) | 36.20 (11.90)
  PCS: Change at Month 6 (n= 18) | 1.60 (7.25)
  PCS: Change at Month 12 (n= 18) | -0.40 (8.47)
  MCS: Baseline (n= 21) | 47.00 (10.96)
  MCS: Change at Month 6 (n= 18) | -1.70 (10.02)
  MCS: Change at Month 12 (n= 18) | 3.00 (11.11)
  Physical functioning: Baseline (n= 21) | 33.20 (14.68)
  Physical functioning: Change at Month 6 (n= 19) | 0.90 (7.50)
  Physical functioning: Change at Month 12 (n= 18) | -0.10 (10.84)
  Role-physical: Baseline (n= 21) | 38.90 (13.80)
  Role-physical: Change at Month 6 (n= 19) | -1.80 (10.42)
  Role-physical: Change at Month 12 (n= 18) | -3.80 (12.91)
  Bodily pain: Baseline (n= 21) | 45.50 (11.27)
  Bodily pain: Change at Month 6 (n= 19) | 0.80 (9.42)
  Bodily pain: Change at Month 12 (n= 18) | 1.50 (10.11)
  General health: Baseline (n= 21) | 36.00 (9.47)
  General health: Change at Month 6 (n= 19) | 2.70 (9.97)
  General health: Change at Month 12 (n= 18) | 4.00 (10.33)
  Vitality: Baseline (n= 21) | 43.30 (11.83)
  Vitality: Change at Month 6 (n= 18) | 1.20 (7.95)
  Vitality: Change at Month 12 (n= 18) | 3.10 (9.93)
  Social functioning: Baseline (n= 21) | 41.80 (11.16)
  Social functioning: Change at Month 6 (n= 19) | 2.00 (11.09)
  Social functioning: Change at Month 12 (n= 18) | 3.00 (11.72)
  Role-emotional: Baseline (n= 21) | 41.60 (14.82)
  Role-emotional: Change at Month 6 (n= 19) | -1.20 (7.45)
  Role-emotional: Change at Month 12 (n= 18) | 0.40 (12.43)
  Mental health: Baseline (n= 21) | 46.90 (10.11)
  Mental health: Change at Month 6 (n= 18) | -3.80 (11.47)
  Mental health: Change at Month 12 (n= 18) | 2.00 (12.44)

18. Other Pre Specified Outcome: Change From Baseline in Echocardiography (ECHO) Parameters at Month 6, Month 12
Description: Echocardiography was used to measure interventricular septal thickness (IVST), posterior left ventricular wall thickness (PLVWT), right ventricular wall thickness (RVWT), left atrial diameter (LAD): anterior-posterior (ant-post), medio-lateral, superior-inferior (sup-inf) and left ventricular end diastolic diameter (LVED), relative LV wall thickness (RLVWT).
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
millimeter (mm)
  IVST: Baseline (n=19) | 15.24 (2.77)
  IVST: Change at Month 6 (n=15) | 0.57 (2.10)
  IVST: Change at Month 12 (n=14) | 1.04 (2.04)
  PLVWT: Baseline (n=19) | 14.60 (2.59)
  PLVWT: Change at Month 6 (n=15) | 0.30 (1.98)
  PLVWT: Change at Month 12 (n=14) | 0.70 (1.73)
  RVWT: Baseline (n=17) | 6.09 (2.01)
  RVWT: Change at Month 6 (n=8) | 1.12 (1.72)
  RVWT: Change at Month 12 (n=12) | 1.08 (1.29)
  LAD (ant-post): Baseline (n=21) | 36.30 (6.20)
  LAD (ant-post): Change at Month 6 (n=17) | 1.50 (4.57)
  LAD (ant-post): Change at Month 12 (n=16) | 1.60 (3.52)
  LAD (medio-lateral): Baseline (n=16) | 37.40 (4.80)
  LAD (medio-lateral): Change at Month 6 (n=7) | 4.30 (6.90)
  LAD (medio-lateral): Change at Month 12 (n=9) | 1.90 (4.20)
  LAD (sup-inf): Baseline (n=16) | 48.30 (9.88)
  LAD (sup-inf): Change at Month 6 (n= 8) | 3.10 (5.03)
  LAD (sup-inf): Change at Month 6 (n= 9) | 4.20 (6.46)
  LVED: Baseline (n= 19) | 39.66 (4.84)
  LVED: Change at Month 6 (n= 15) | -1.03 (3.88)
  LVED: Change at Month 12 (n= 14) | 0.11 (3.42)
  RLVWT: Baseline (n=19) | 0.75 (0.19)
  RLVWT: Change at Month 6 (n= 15) | 0.05 (0.16)
  RLVWT: Change at Month 12 (n= 14) | 0.03 (0.12)

19. Other Pre Specified Outcome: Change From Baseline in Left Atrial Volume at Month 6, Month 12
Description: Left atrial volume was measured by echocardiography.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: cubic centimeter (cc)
Arm/Group | Tafamidis
Number analyzed (Participants) | 15
cubic centimeter (cc)
  Baseline (n= 15) | 51.50 (23.81)
  Change at Month 6 (n= 6) | 12.30 (17.20)
  Change at Month 12 (n= 9) | 1.90 (18.90)

20. Other Pre Specified Outcome: Change From Baseline in Left Ventricular (LV) End Systolic Volume, Left Ventricle (LV) Stroke Volume at Month 6, Month 12
Description: Cardiac MRI was done to measure left ventricular (LV) end systolic volume, left ventricle (LV) stroke volume.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Tafamidis
Number analyzed (Participants) | 11
milliliter (mL)
  LV end systolic volume: Baseline (n= 11) | 30.4 (13.93)
  LV end systolic volume: Change at Month 6 (n= 6) | 3.50 (7.79)
  LV end systolic volume: Change at Month 12 (n= 6) | 4.70 (3.01)
  LV stroke volume: Baseline (n= 11) | 43.10 (13.26)
  LV stroke volume: Change at Month 6 (n= 6) | -2.50 (15.23)
  LV stroke volume: Change at Month 12 (n= 6) | 3.70 (10.69)

21. Other Pre Specified Outcome: Change From Baseline in Fractional Shortening at Month 6, Month 12
Description: Fractional shortening (FS) is the fraction of any diastolic dimension that is lost in systole. Percent of FS was calculated as difference between end-diastolic dimension (EDD) and end-systolic dimension (EDS) divided by EDD.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of EDD
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
percentage of EDD
  Baseline (n= 18) | 31.20 (5.68)
  Change at Month 6 (n= 14) | -1.10 (5.91)
  Change at Month 12 (n= 14) | -0.90 (6.24)

22. Other Pre Specified Outcome: Change From Baseline in Left Ventricular (LV) Ejection Fraction at Month 6, Month 12
Description: Cardiac MRI was done to measure left ventricular ejection fraction (LVEF) which was the fraction of the end-diastolic volume (EDV) that was ejected out of left ventricle with each contraction.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of EDV
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
percentage of EDV
  Baseline (n= 21) | 60.30 (9.96)
  Change at Month 6 (n= 18) | -3.80 (7.73)
  Change at Month 12 (n=18) | -2.20 (5.37)

23. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Mass (LVM) at Month 6, Month 12
Description: LV mass was calculated from the product of the myocardial volume and specific gravity of heart muscle, estimated by echocardiography. Increased LVM was associated with cardiovascular morbidity and mortality.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Tafamidis
Number analyzed (Participants) | 19
gram
  Baseline: (n= 19) | 230.84 (62.54)
  Change at Month 6 (n= 15) | 1.11 (46.53)
  Change at Month 12 (n= 14) | 20.91 (35.07)

24. Other Pre Specified Outcome: Change From Baseline in Isovolumetric Relaxation Time (IVRT), Mitral Deceleration Time at Month 6, Month 12
Description: Doppler echocardiography was a procedure which used ultrasound technology to examine the heart. IVRT is the time between the closure of the aortic valve and the opening of the mitral valve. Mitral deceleration time (MDT) was the time taken from the maximum E point wave to baseline. E wave arises due to early diastolic filling.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
msec
  IVRT: Baseline (n= 10) | 84.10 (17.51)
  IVRT: Change at Month 6 (n= 3) | 2.70 (20.03)
  IVRT: Change at Month 12 (n= 8) | -4.00 (25.63)
  MDT: Baseline (n= 18) | 164.00 (35.59)
  MDT: Change at Month 6 (n= 14) | 1.90 (28.17)
  MDT: Change at Month 12 (n= 15) | 11.90 (29.45)

25. Other Pre Specified Outcome: Change From Baseline in Aortic Annulus Diameter at Month 6, Month 12
Description: The diameter at the base of the aortic root, the basal ring, is also called the aortic annulus diameter.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
centimeter (cm)
  Baseline (n= 21) | 2.045 (0.184)
  Change at Month 6 (n= 17) | -0.009 (0.160)
  Change at Month 12 (n= 16) | -0.041 (0.108)

26. Other Pre Specified Outcome: Change From Baseline in Tricuspid Peak Velocity at Month 6, Month 12
Description: Tricuspid peak velocity was measured by echocardiography.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: meter per second (m/sec)
Arm/Group | Tafamidis
Number analyzed (Participants) | 11
meter per second (m/sec)
  Baseline (n= 11) | 26.80 (8.62)
  Change at Month 6 (n= 9) | 0.90 (4.86)
  Change at Month 12 (n= 8) | 2.10 (9.25)

27. Other Pre Specified Outcome: Change From Baseline in Tricuspid Pulmonary Artery Systolic Pressure (PASP) at Month 6, Month 12
Description: Systolic right ventricular pressure can be estimated on echocardiography by adding right atrial pressure (RAP) to the trans-tricuspid gradient derived from the tricuspid regurgitation velocity.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Tafamidis
Number analyzed (Participants) | 11
millimeter of mercury (mmHg)
  Baseline (n= 11) | 35.50 (11.55)
  Change at Month 6 (n= 6) | 3.80 (7.81)
  Change at Month 12 (n= 7) | 2.10 (13.08)

28. Other Pre Specified Outcome: Change From Baseline in Doppler Data at Month 6, Month 12
Description: Doppler echocardiography was a procedure which used ultrasound technology to examine the heart. Doppler principle was used to measure the mitral peak early (E) diastolic transmitral flow, mitral peak atrial (A) contraction velocity and annular velocities at the lateral and septal areas of the mitral annulus. s': systolic velocity during ejection, e': early diastolic mitral annular velocity, a': late diastolic mitral annular velocity.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: centimeter per second (cm/sec)
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
centimeter per second (cm/sec)
  Mitral Peak A: Baseline (n= 18) | 59.00 (23.77)
  Mitral Peak A: Change at Month 6 (n= 13) | -0.50 (16.01)
  Mitral Peak A: Change at Month 12 (n= 15) | -3.70 (15.43)
  Mitral Peak E: Baseline (n= 19) | 74.10 (15.58)
  Mitral Peak E: Change at Month 6 (n= 15) | 4.70 (10.28)
  Mitral Peak E: Change at Month 12 (n= 16) | 5.10 (13.75)
  Septal s': Baseline (n= 16) | 4.72 (1.64)
  Septal s': Change at Month 6 (n= 12) | 0.43 (0.51)
  Septal s': Change at Month 12 (n= 8) | -0.33 (0.90)
  Septal e': Baseline (n= 16) | 4.54 (1.88)
  Septal e': Change at Month 6 (n= 12) | 1.25 (2.29)
  Septal e': Change at Month 12 (n= 8) | 0.04 (0.61)
  Septal a': Baseline (n= 15) | 4.66 (2.67)
  Septal a': Change at Month 6 (n= 11) | 0.53 (1.39)
  Septal a': Change at Month 12 (n= 8) | -0.10 (1.74)
  Lateral s': Baseline (n= 16) | 6.71 (2.97)
  Lateral s': Change at Month 6 (n= 10) | 0.55 (1.41)
  Lateral s': Change at Month 12 (n= 7) | 0.19 (1.20)
  Lateral e': Baseline (n= 16) | 6.91 (2.90)
  Lateral e': Change at Month 6 (n= 11) | 0.65 (1.27)
  Lateral e': Change at Month 12 (n= 7) | 0.16 (1.42)
  Lateral a': Baseline (n= 15) | 5.93 (3.38)
  Lateral a': Change at Month 6 (n= 10) | 0.31 (2.69)
  Lateral a': Change at Month 12 (n= 6) | -0.45 (2.94)

29. Other Pre Specified Outcome: Change From Baseline in e:e' Lateral Ratio , Ratio of Peak Mitral Early Diastolic and Atrial Contraction Velocity (E/A Ratio) at Month 6, Month 12
Description: Doppler echocardiography was a procedure which used ultrasound technology to examine the heart. Ratio of early (E) diastolic transmitral flow velocity and atrial (A) contraction velocity (E/A) and ratio of the early (E) diastolic transmitral flow velocity to the mitral annular velocity (e') (E/e') were estimated.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
ratio
  e:e' Lateral: Baseline (n= 16) | 13.148 (7.781)
  e:e' Lateral: Change at Month 6 (n= 10) | -0.145 (3.227)
  e:e' Lateral: Change at Month 12 (n= 7) | -0.243 (5.245)
  E/A: Baseline (n= 18) | 1.463 (0.667)
  E/A: Change at Month 6 (n= 13) | 0.175 (0.565)
  E/A: Change at Month 12 (n= 15) | 0.185 (0.658)

30. Other Pre Specified Outcome: Change From Baseline in Left Ventricular (LV) Mass/Voltage Ratio at Month 6, Month 12
Description: LV mass was calculated from the product of the myocardial volume and specific gravity of heart muscle, estimated by echocardiography. QRS score (the sum of QRS voltages in the peripheral leads) was used as an index of "electrical" LV mass.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: gram/millivolt
Arm/Group | Tafamidis
Number analyzed (Participants) | 19
gram/millivolt
  Baseline (n= 19) | 5.495 (2.149)
  Change at Month 6 (n= 14) | 0.028 (1.479)
  Change at Month 12 (n= 14) | 0.878 (1.437)

31. Other Pre Specified Outcome: Change From Baseline in Left Atrial (LA) Volume Index at Month 6, Month 12
Description: LA volume index (LAVI), was the value of LA volume divided by body surface area, to measure LA size.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliliter/square meter (mL/m^2)
Arm/Group | Tafamidis
Number analyzed (Participants) | 15
milliliter/square meter (mL/m^2)
  Baseline (n= 15) | 27.33 (10.21)
  Change at Month 6 (n= 5) | 7.23 (8.78)
  Change at Month 12 (n= 9) | 1.06 (9.66)

32. Other Pre Specified Outcome: Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) at Week 2, Week 6, Month 3, Month 6, Month 12
Description: NT-proBNP was a cardiac marker which had the prognostic value for participants with heart failure or left ventricular dysfunction. Higher level of the marker was indicative of heart damage.
Time Frame: Baseline, Week 2, Week 6, Month 3, Month 6, Month 12
Population: ITT population. Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were analyzed for the specific category. Data prior Month 6 were not anticipated to be informative hence were not analyzed.
Measure: Mean (Standard Deviation); unit: picogram/mL (pg/mL)
Arm/Group | Tafamidis
Number analyzed (Participants) | 19
picogram/mL (pg/mL)
  Baseline (n= 19) | 1248.89 (1529.37)
  Change at Month 6 (n= 18) | 228.39 (834.91)
  Change at Month 12 (n= 16) | 306.61 (1447.67)

33. Other Pre Specified Outcome: Change From Baseline in Karnofsky Performance Status Scale at Month 6, Month 12
Description: Karnofsky performance score is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. Karnofsky performance score is 11 level score which ranges between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 21
units on a scale
  Baseline (n= 21) | 74.80 (14.01)
  Change at Month 6 (n= 19) | -1.10 (5.67)
  Change at Month 12 (n= 18) | -3.30 (5.94)

34. Other Pre Specified Outcome: Change From Baseline in Troponin I Levels at Week 2, Week 6 , Month 3, Month 6, Month 12
Description: Troponin I is a cardiac injury biomarker. Higher concentrations of this marker in blood are associated with heart injury.
Time Frame: Baseline, Week 2, Week 6 , Month 3, Month 6, Month 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: nanogram/mL
Arm/Group | Tafamidis
Number analyzed (Participants) | 20
nanogram/mL
  Baseline (n= 20) | 0.0234 (0.0409)
  Change at Month 6 (n= 18) | 0.0015 (0.0501)
  Change at Month 12 (n= 18) | 0.0025 (0.0487)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tafamidis
Serious Adverse Events (participants affected / at risk) | 8/21
Other Adverse Events (participants affected / at risk) | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis (N=21)
Atrioventricular block (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis (N=21)
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 2
Laryngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Neuralgia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.